## An Investigation of the Physical Task Demands of Caregivers Working in a Long-Term Care Facility

Study Protocol and Appendix

Dubé A<sup>1</sup>., Brun C<sup>1</sup>., Albert WJ<sup>2</sup>. & Cardoso MR<sup>1</sup>.

Université de Moncton University of New Brunswick

May 29th, 2024

#### **Appendix A: Ergonomic Tool**

| Participant ID: | No: |
|-----------------|-----------|
| Data | Lagation |
| Date: | Location: |

The aim of the evaluation is to observe and record the various motor tasks performed by the participants during a typical day at work.

There will be no assessment of movement quality or techniques used; the aim is simply to count and record the number of times each movement or motor task has been performed during the day.

#### **Part 1: Patient Transfers**

A- The caregiver did NOT use any tools or aids while performing the following transfer tasks:

| Type of transfers requiring Physical assistance from the caregiver | Number of transfers completed | Resident condition 1. No assistance from resident 2. Assist/Help 3. Guidance only | Duration<br>(minutes):<br>Record 3<br>separate trials |
|---|---|---|---|
| Bed to Wheelchair | | | AM 1 - 2 - 3 - PM 1 - 2 - 3 - 3 - |
| Wheelchair to Bed | | | AM 1 - 2 - 3 - PM 1 - 2 - 3 - 3 - |
| Wheelchair to chair | | | AM<br>1 -<br>2 -<br>3 - |

| | 1 - 2 - 3 - | PM |
|----------------------|-------------------|----------|
| Chair to Wheelchair | 1 –<br>2 –<br>3 – | AM<br>PM |
| Wheelchair to Toilet | 1 –<br>2 –<br>3 – | AM<br>PM |
| Toilet to Wheelchair | 1 –<br>2 –<br>3 – | AM<br>PM |

# B- The caregiver used tools and/or aids while performing the following transfer tasks:

| Type of transfers requiring physical assistance from the caregiver | Number of transfers completed | Resident condition 1. No assistance from resident 2. Assist/Help 3. Guidance only | Duration<br>(minutes):<br>Record 3<br>separate trials |
|---|---|---|---|
| Bed to Wheelchair – with the use of tools/aids | | | AM<br>1 -<br>2 -<br>3 - |
| | | | PM<br>1 -<br>2 -<br>3 - |
| Wheelchair to Bed – with the use of tools/aids | | | AM 1- 2- 3- |
| | | | PM<br>1 –<br>2 –<br>3 – |
| Wheelchair to Chair – with the use of tools/aids | | | AM<br>1 –<br>2 –<br>3 – |
| | | | PM<br>1 -<br>2 -<br>3 - |
| Chair to Wheelchair – with the use of tools/aids | | | AM<br>1 -<br>2 -<br>3 - |

| | PM<br>1 -<br>2 -<br>3 - |
|---|---|
| Wheelchair to Toilet – with the use of tools/aids | AM 1 - 2 - 3 - PM 1 - 2 - 3 - 3 - |
| Toilet to Wheelchair – with the use of tools/aids | AM 1 - 2 - 3 - PM 1 - 2 - 3 - 3 - |

C- Tools used by caregiver for resident transfers:

| Type of tool <u>used with mechanical assistance</u> when transferring the resident (e.g., ceiling | Number of transfers completed |
|---|---|
| lifts). | |
| Type of tool used WITHOUT mechanical | Number of transfers completed |
| Type of tool <u>used WITHOUT mechanical</u> <u>assistance</u> when transferring the resident (e.g., transfer boards). | Number of transfers completed |
| <u>assistance</u> when transferring the resident (e.g., | Number of transfers completed |

# Part 2: Resident handling A - Resident handling in <u>Bed</u>

| <b>Resident handling Movement Patterns</b> | Number of handlings completed |
|---|---|
| Side to side (turning a resident to their side ex: Turn 1, Turn 2) | |
| Straightening (sit/back) | |
| Side bearing | |
| Pull a patient up in bed (ex: Up in Bed) (vertical) | |
| Pull a patient down in bed (ex: Up in Bed) (vertical) | |
| Horizontal pull (ex: Side 1, Side 2) | |
| Horizontal pull (lower limbs) | |
| Additional Movement Patterns | |

## B: Resident handling in Wheelchair - Sitting

| Motor task | Number of handlings completed |
|-------------------------------------|-------------------------------|
| Side to side | |
| Lift up | |
| Repositioning of lower limbs | |
| responding of lower miles | |
| <b>Additional Movement Patterns</b> | |

## Part 3: Motor tasks – Housework – Sanitary

| Motor tasks | Number of times completed |
|-------------------------------------------------|---------------------------|
| Making a bed | |
| Leaning towards the ground (e.g., picking | |
| up an object, rubbing dirt on the floor) | |
| Lifting an object that weighing more than | |
| 10 pounds | |
| 1 | |
| A selection of a month of and the first and the | |
| Assisting the resident with their bathing needs | |
| needs | |
| Washing a resident independently | |
| (without help) | |
| Assisting a resident to walk | |
| Assisting in dressing and undressing a | |
| resident | |
| Assisting a resident to eat | Standing: |
| Tissisting a resident to ear | Sumonig. |
| | Sitting: |
| Other | |

Part 4: Time spent under different type of behaviors (lasting more than 10 mins)

| Workplace Movement | Number of times (+10mins) | Duration (minutes):<br>Record 3 separate<br>trials |
|---|---|---|
| Standing (working) | | 1 –<br>2 –<br>3 – |
| Sitting (working) | | 1 –<br>2 –<br>3 – |
| Walking (working) | | 1 –<br>2 –<br>3 – |
| Walking (pushing a wheelchair or carrying an object) - loading | | 1 –<br>2 –<br>3 – |
| Other | | |
| | | 1 - 2 - 3 - |

#### Part 5: Additional Information

| Number of hours worked without a break |
|----------------------------------------|
| (max) |
| Total hours worked |
| Total rest time (hours) |
| Other |

Part 6: Field observations:

#### **APPENDIX B – Rate of Perceived Questionnaire (RPD)**

## Patient handling







## Appendix C: H&L-Q (Lifestyle Questionnaire)

| Partic | ipant ID | Date | |
|---|---|---|---|
| Sex | Age | Years of experience in the field | |
| Work | status (full-time or par | rt-time): | |
| Answe | er the next section to t | he best of your knowledge. | |
| | How many times per | week do you participate in cardiovascupgging, biking, swimming; etc.) | |
| | | verage)minutes. Total: | |
| 2. | exercise (lifting weigh | week do you participate in strength trants, body weight exercises, bands; etc.) verage)minutes. Total: | |
| 3. | How many average u oz/week. | nits of alcohol (1oz) do you consume po | er week? |
| 4. | , . | pacco user? If so, do you consume daily<br>few times a week? (Yes or No) | ? (Yes or No) Or, do |
| | What form of tobacco | o do you use? (Cigarette, Vape, Chew, o | or Other) |
| 5. | poor and 10 being gr | your average quality of sleep on a scale eat)? bedtime and wake up schedule? | |
| How r | nuch time do you sper | nd in a sedentary behavior at <b>home</b> (ex: | sitting, laying down |
| | . • • | | |

screentime...)

- 1) Less than 2 hours/day
- 2) Between 2 to 4 hours/day
- 3) Between 4 to 6 hours/day
- 4) Between 6 to 8 hours/day
- 5) More than 8 hours/day

How much time do you spend in a sedentary behavior at **work** (ex: sitting, laying down screentime...)

- 1) Less than 2 hours/day
- 2) Between 2 to 4 hours/day
- 3) Between 4 to 6 hours/day
- 4) Between 6 to 8 hours/day
- 5) More than 8 hours/day

Have you ever experienced work-related musculoskeletal injury (muscle, ligament or bone injuries that affect your ability to perform your job or interfere with your everyday life)

- 1. Yes
- 2. No

If yes, please fill out this Nordic questionnaire:

**Important note**: The term "discomfort" refers to persistent discomfort caused by musculoskeletal injury or pain, and the terms "tightness" or "stiffness" that are **NOT** persistent are not applicable to this term.

| | | Have you at any<br>time during the last<br>12 months had<br>trouble (such as<br>ache, pain,<br>discomfort,<br>numbness) in: | | During the last 12 months<br>have you been prevented<br>from carrying out normal<br>activities (e.g. job,<br>housework, hobbies)<br>because of this trouble in: | | During the last 12<br>months have you<br>seen a physician for<br>this condition: | | During the last 7<br>days have you had<br>trouble in: | |
|---|---|---|---|---|---|---|---|---|---|
| | NECK | □No | Yes | □No | Yes | □No | Yes | □No | Yes |
| | SHOULDERS | □ No | Yes | □No | ☐ Yes | □No | ☐ Yes | □No | ☐ Yes |
| | UPPER BACK | □ No | ☐ Yes | □No | ☐ Yes | □No | ☐ Yes | □No | ☐ Yes |
| | ELBOWS | □No | ☐ Yes | □ No | Yes | □No | Yes | □No | ☐ Yes |
| | WRISTS/ HANDS | □ No | ☐ Yes | □No | Yes | □No | ☐ Yes | □No | ☐ Yes |
| | SOWER BACK | □No | Yes | □ No | Yes | □No | ☐ Yes | □No | ☐ Yes |
| | HIPS/ THIGHS | □ No | Yes | □ No | Yes | □No | ☐ Yes | □ No | ☐ Yes |
| | KNEES | □No | Yes | □ No | Yes | □No | ☐ Yes | □ No | ☐ Yes |
| \$ \$ | ANKLES/ FEET | □ No | Yes | □ No | ☐Yes | □ No | ☐ Yes | □ No | ☐ Yes |

| If yes, how, and when did the injury (ies) occurred. |
|---|
| ; |
| Did you have to take some time off from work due to this injury, if so, please elaborate: |
| How would you rate the overall physical demands of your work? 1. Very Easy 2. Easy 3. Average 4. Difficult 5. Very Difficult |
| Based on your baseline level at the start of the day, how would you rate your level of fatigue at the end of your workday on average on a scale of 0 to 10? |
| What suggestions do you have for interventions or strategies that could potentially reduce the physical demands of your work and ensure your safety and well-being at work? |
| General Comments: |